CLINICAL TRIAL: NCT00269841
Title: A Placebo-Controlled, Repeated-Dose Study of Anti-TNF Chimeric Monoclonal Antibody (cA2) in the Treatment of Patients With Enterocutaneous Fistulae as a Complication of Crohn's Disease
Brief Title: An Efficacy and Safety Study of Anti-TNF Monoclonal Antibody in Patients With Fistulizing Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006253
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Crohn Disease
Keywords: fistulae; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Infliximab 10 mg/kg (Experimental): Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 10 milligram per kilogram (mg/kg) will be administered as infusion at Week 0, 2 and 6.
  Interventions: Drug: Infliximab 10 mg/kg
- Infliximab 5 mg/kg (Experimental): Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 5 mg/kg will be administered as infusion at Week 0, 2 and 6.
  Interventions: Drug: Infliximab 5 mg/kg
- Placebo (Placebo Comparator): Matching placebo will be administered at Week 0, 2 and 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab 10 mg/kg — Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 10 milligram per kilogram (mg/kg) will be administered as infusion at Week 0, 2 and 6.
  Other Names: anti-TNF chimeric monoclonal antibody (cA2)
  Arms: Infliximab 10 mg/kg
Drug: Infliximab 5 mg/kg — Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 5 mg/kg will be administered as infusion at Week 0, 2 and 6.
  Other Names: anti-TNF chimeric monoclonal antibody (cA2)
  Arms: Infliximab 5 mg/kg
Drug: Placebo — Matching placebo will be adminstered at Week 0, 2 and 6.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of anti-TNF chimeric monoclonal antibody (cA2) compared to placebo in the treatment of patients with fistulizing Crohn's disease.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, repeated-dose study to evaluate the effectiveness and safety of anti-TNF chimeric monoclonal antibody (cA2) compared to placebo in the treatment of patients with fistulizing Crohn's disease. The primary efficacy outcome of the study is the number of patients with at least a 50% reduction from baseline in the number of open fistulae observed for at least two consecutive evaluation visits.

Patients will be treated with either anti-TNF chimeric monoclonal antibody (cA2) or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease of at least 3 months duration confirmed by radiography orendoscopy
* Having single or multiple draining enterocutaneous (including perianal) fistulae of at least 3 months duration
* If treated with oral prednisone (or equivalent), the dose must be <=40 mg/day and must have been stable for at least 3 weeks prior to enrollment. (If currently not treated with oral prednisone, the stop date must have been at least 4 weeks prior to enrollment)
* If treated with 6-mercaptopurine or azathioprine, the start date must have been at least 6 months prior to enrollment. (The dose must have been stable for at least 8 weeks prior to enrollment. If currently not treated with 6-mercaptopurine or azathioprine, the stop date must have been at least 4 weeks prior to enrollment.)

Exclusion Criteria:

* Patients with local complications of Crohn's disease such as strictures or abscesses that might confound the evaluations of the benefit from cA2 treatment
* Having abscesses that should be drained prior to enrollment, with at least 3 weeks between drainage of the abscess and enrollment
* Having a serious infection, such as hepatitis, pneumonia or pyelonephritis, in the previous 3 months or a history of opportunistic infection such as herpes zoster within 2 months prior to screening, or evidence of active cytomegalovirus, active pneumocystis carinii, or drug resistant atypical mycobacterium
* Currently having signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease
* Currently having any known malignancy or any history of malignancy within the past 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 1996-05; Primary Completion 1998-02 (Actual); Study Completion 1998-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with 50% or more reduction from baseline in the number of open fistulae at Week 3 | Week 3
  Number patients with 50% or more reduction from baseline in the number of open fistulae observed for at least two consecutive evaluation visits that is not accompanied by initiation of a therapeutic agent or increase in dose.

SECONDARY OUTCOMES:
Percentage of patients achieving a complete response at week 52 | Week 52
  The percentage of patients achieving a complete response; In patients responding to treatment, the median time to first observed reduction from baseline of 50% or greater in the number of open fistulae

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Present DH, Rutgeerts P, Targan S, Hanauer SB, Mayer L, van Hogezand RA, Podolsky DK, Sands BE, Braakman T, DeWoody KL, Schaible TF, van Deventer SJ. Infliximab for the treatment of fistulas in patients with Crohn's disease. N Engl J Med. 1999 May 6;340(18):1398-405. doi: 10.1056/NEJM199905063401804. PMID 10228190